CLINICAL TRIAL: NCT02337309
Title: Phase I Study of SF1126 for Patients With Relapsed or Refractory Neuroblastoma
Brief Title: SF1126 for Patients With Relapsed or Refractory Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low patient accrual
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: SignalRX Pharmaceuticals, Inc. (Industry); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NANT 2014-01; N14-01 (Other: NANT Consortium); R01FD005740 (FDA)
Record Dates: First submitted 2014-12-18; First posted 2015-01-13 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — SF 1126

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SF1126 (Other): Patients will receive SF1126 IV over 90 minutes on Days 1 and 4 of each week during each cycle.
  Interventions: Drug: SF1126

INTERVENTIONS:
Drug: SF1126 — SF1126 in IV form with be given to patients on this study.

SUMMARY:
SF1126 is a novel inhibitor of PI3 kinase and mTOR that includes an active moiety (consisting of LY294002) linked to an RGDS tetrapeptide that targets the active agent to integrin expressing tissues. In this first pediatric phase 1 trial of SF1126, dose escalation will follow a 3+3 dose escalation design. Once a recommended phase 2 pediatric dose is identified, an expansion cohort of 10 patients with tumors with MYCN amplification, Mycn expression, or Myc expression will be treated.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Inhibitors of the PI3 kinase pathway have demonstrated preclinical activity in neuroblastoma. This activity may derive in part from destabilizing Mycn protein, impeding tumor angiogenesis, and/or other effects. SF1126 is a novel inhibitor of PI3 kinase and mTOR that includes an active moiety (consisting of LY294002) linked to an RGDS tetrapeptide that targets the active agent to integrin expressing tissues. In preclinical studies, SF1126 results in marked concentration of LY294002 into tumors. In an adult phase 1 trial, a maximum tolerated dose of SF1126 was not identified up to doses of 1110 mg/m2 administered intravenously twice weekly on a continuous schedule. In this first pediatric phase 1 trial of SF1126, dose escalation will follow a 3+3 dose escalation design. Once a recommended phase 2 pediatric dose is identified, an expansion cohort of 10 patients with tumors with MYCN amplification, Mycn expression, or Myc expression will be treated. All patients will participate in mandatory pharmacokinetic testing. Additional optional correlative studies will evaluate potential predictive markers and potential pharmacodynamic markers, including PTEN and PIK3CA aberrations, Myc / Mycn expression, and Myc / pS6 levels in peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
* Patients must have high-risk neuroblastoma according to COG risk classification at the time of study enrollment.
* Patients must have at least ONE of the following: 1) Recurrent/progressive disease at any time prior to study enrollment, 2) Refractory disease, 3) Persistent disease
* Patients must have at least ONE of the following: 1) Bone disease, 2) Any amount of neuroblastoma tumor cells in the bone marrow, 3) At least one soft tissue lesion that meets criteria for a TARGET lesion.
* Patients must have a Lansky (< 16 years) or Karnofsky (> 16 years) score of at least 50
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Patients must not be receiving any other anti-cancer agents or radiotherapy at the time of study entry or while on study.
* Patients must not be receiving other investigational medications (covered under another IND) within 30 days of study entry or while on study.
* Patients must not be receiving chronic systemic corticosteroids at doses greater than physiologic dosing (inhaled corticosteroids acceptable).
* Patient must meet the organ function requirements as stated in the protocol.

Exclusion Criteria:

* Pregnancy, breast feeding, or unwillingness to use effective contraception during the study.
* Patients status post-allogeneic stem cell transplant are not eligible.
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
* Patients with disease of any major organ system that would compromise their ability to withstand therapy.
* Patients who are on hemodialysis.
* Patients with an active or uncontrolled infection.
* Patients with known intraparenchymal brain metastasis at study entry are excluded due to poor CNS penetration of SF1126.
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C.
* Patient declines participation in NANT 2004-05, the NANT Biology Study.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Toxicities, based on the CTCAE criteria, will be used to measure the severity of adverse events | 6 months
  Toxicity will be graded using the CTCAE criteria, version 4. The CTCAE provides descriptive terminology and a grading scale for each adverse event listed. A copy of the CTCAE can be downloaded from the CTEP home page (http://ctep.cancer.gov).

SECONDARY OUTCOMES:
Evaluation of response | After day 1 of week 4 of cycles 2, 4, and 6
  Response will be determined by the evaluation of CT/MRI scans and bone marrow biopsy.
Pharmacokinetics: Parameters include AUC, clearance, Cmax, Tmax, & terminal half-life for SF1101 & SF1174. With rapid conversion of SF1126 to SF1101, only AUC, clearance, Cmax & Tmax are calculated for SF1126. | Day 1, cycle 1
  Plasma samples will be collected from patients at 9 time points on Day 1 of the first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Steven DuBois, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Childrens Hospital Boston, Dana-Farber Cancer Institute., Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cook Children's Healthcare System, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No